CLINICAL TRIAL: NCT07283952
Title: Diverting Ileostomy Verses Transverse Colostomy in Colorectal Surgery
Brief Title: Diverting Ileostomy and Transverse Colostomy Comparative Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Esam Ahmed Taher Mahmoud, Resident at the Department of General Surgery, Assiut University, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Stoma Type Comparison
Record Dates: First submitted 2025-11-20; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-11

CONDITIONS: Ileostomy; Colostomy; Colorectal Surgery
Keywords: Diverting Ileostomy; Transverse Colostomy; Colorectal Surgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- diverting ileostomy (Active Comparator)
  Interventions: Procedure: Diverting ileostomy
- transverse colostomy (Active Comparator)
  Interventions: Procedure: Diverting Transverse Colostomy

INTERVENTIONS:
Procedure: Diverting ileostomy — a surgical procedure in which the a segment of the ileum is mobilized and placed as a stoma diverting technique to protect any distal anastomosis
  Arms: diverting ileostomy
Procedure: Diverting Transverse Colostomy — a surgical procedure in which the a segment of the transverse colon is mobilized and placed as a stoma diverting technique to protect any distal anastomosis.
  Arms: transverse colostomy

SUMMARY:
Protective diverting stomas are frequently constructed after low anterior resection or colorectal anastomosis to mitigate the consequences of anastomotic leakage, one of the most feared complications in colorectal surgery.

Both loop ileostomy (LI) and loop transverse colostomy (TC) are accepted methods of diversion. Randomized and observational studies have shown that faecal diversion significantly reduces the clinical severity of leaks and the need for reoperation compared with no diversion.

The choice between LI and TC remains controversial. Loop ileostomy is technically straightforward and associated with shorter operative time and fewer septic complications at closure. However, it carries specific risks, including high-output stoma, dehydration, electrolyte imbalance, and renal impairment, which may lead to hospital readmissions. Conversely, loop transverse colostomy is associated with fewer fluid and electrolyte issues, but has higher rates of prolapse, skin irritation, and wound complications at closure.

Meta-analyses comparing LI and TC indicate no clear superiority, with each approach demonstrating distinct patterns of morbidity. Some randomized trials have suggested lower major morbidity with LI, while others found no significant difference. Given the heterogeneity of outcomes and limited high-quality, adequately powered trials, further randomized evidence is needed to guide optimal stoma selection in colorectal surgery.

ELIGIBILITY:
Inclusion Criteria:

* • Adults ≥18 years undergoing elective low anterior resection or coloanal anastomosis for benign or malignant colorectal disease.

  * Patients for whom the surgeon has decided that a diverting stoma is required such as emergency resection and anastomosis cases where a covering stoma is indicated.
  * Ability to provide informed consent.

Exclusion Criteria:

* • Patients with pre-existing stoma.

  * Severe comorbidities precluding stoma creation (e.g., advanced renal failure, uncontrolled cardiac disease).
  * Patients with extensive peritoneal carcinomatosis or unresectable disease.
  * Pregnant or lactating women.
  * Inability to comply with follow-up or provide informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Clinically or Radiologically Confirmed Anastomotic Leak | From index colorectal surgery to 30 days after surgery
  Count of participants in each arm who develop an anastomotic leak confirmed by clinical signs (such as fever, abdominal pain, peritonitis, or purulent discharge) and/or by contrast-enhanced radiological imaging. The unit of measure will be number of participants.
Severity of Anastomotic Leak Assessed by Clavien-Dindo Classification | From index colorectal surgery to 30 days after surgery
  Distribution of Clavien-Dindo complication grades among participants who develop an anastomotic leak in each arm. The unit of measure will be number of participants in each Clavien-Dindo grade category.
Number of Participants With Anastomotic Leak Requiring Surgical Management | From index colorectal surgery to 30 days after surgery
  Count of participants with anastomotic leak who require operative intervention, including re-laparotomy, laparoscopic washout, stoma revision, or creation of a new stoma. The unit of measure will be number of participants.

SECONDARY OUTCOMES:
Intraoperative Blood Loss During Index Surgery | Intraoperative period of index surgery
  Estimated volume of blood loss during the index colorectal resection and stoma creation, as recorded in the anesthesia or operative record. The unit of measure will be milliliters.
Number of Participants With Postoperative Bleeding Requiring Transfusion or Intervention | From index colorectal surgery to 30 days after surgery
  Count of participants who experience postoperative bleeding after index surgery that requires blood transfusion, endoscopic hemostasis, radiological embolization, or reoperation. The unit of measure will be number of participants.
Operative Time for Index Surgery | Intraoperative period of index surgery
  Duration of the index colorectal resection and diverting stoma creation measured from skin incision to skin closure. The unit of measure will be minutes.
Length of Hospital Stay After Index Surgery | Baseline
  Duration of hospitalization in days for the admission during which the index colorectal surgery and stoma creation are performed, from the day of operation to the day of discharge. The unit of measure will be days.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed H Othman, Doctorate, Study Chair — Assiut University; Mohamed abulfetouh, Doctorate, Study Director — Assiut University; Ahmed G Hemdan, doctorate, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Yes
age, brief medical and surgical history , lab investigations and any imaging done pre or post operative
Supporting Information: Study Protocol, CSR